CLINICAL TRIAL: NCT05709639
Title: Exploring the Association of Sport Nutrition Knowledge and Self-reported Physique Concerns on Eating Behaviours in Elite Athletes Receiving Individualized Sport Nutrition Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: Institut National du Sport du Quebec (Unknown); University of Sydney (Other); McMaster University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-08-103
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior | interventions — Nutritional Status; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Responder (Experimental): Increased carbohydrate intake (top 50%) vs moderate to regression in carbohydrate intake (lower 50%)
  Interventions: Other: Individualized counselling in nutrition

INTERVENTIONS:
Other: Individualized counselling in nutrition — Individualized counselling in nutrition - collaborate on a nutrition plan
  Other Names: Nutrition Intervention

SUMMARY:
The Relative Energy Deficiency in Sport (RED-S) syndrome is common in high performance sports, and it impairs athletes' performance and health. The condition is caused by low energy availability (LEA). This means that the body does not have enough energy, after fuelling exercise, to support normal body functions. LEA weakens the structure of bone tissue and increases the risk of bone injuries, lowers your immune function, and increases risk of illnesses, lowers your metabolism, reduces reproductive hormones, and impairs muscle function.

More people are investigating the use of nutrition education programs and individualized nutrition support to improve nutrition knowledge and eating habits in elite athletes. Because the results from available studies look promising, more professionals are examining the effectiveness of different nutrition intervention strategies to improve energy and nutrient intake in athletes. At this point, we do not know if athletes who have higher nutrition knowledge have better eating habits to lower the risk of LEA. Moreover, we do not know what nutrition interventions are useful to improve food intake in athletes who do not eat enough calories for exercise.

With this study we hope to learn if individualized counselling in sport nutrition is associated with changes in eating habits and sport nutrition knowledge in elite athletes to enhance energy availability. It will also teach us if other factors are important to consider when relying on individualized sport nutrition counselling to lower the risk of LEA.

Main Aim: Investigate the differences in individualized nutrition counselling characteristics, sport nutrition knowledge and self-reported body weight and shape concerns between high and low eating behaviour change responders among tier 4 and 5 elite athletes.

Hypothesis: It is hypothesized that self-reported body weight and shape concerns will be negatively associated, and nutrition knowledge will be positively associated with changes in energy and carbohydrate intake in athletes receiving individualized nutrition counselling for 12 weeks.

DETAILED DESCRIPTION:
The aim is to recruit 28 tier 4 and 5 elite athletes through the Canadian Olympic and Paralympic Sport Institute Network and National Sport Organizations between June 2023 and April 2024. Participants will be eligible for inclusion if they compete internationally for Canada at a sport event hosted by an International Federation on the Olympic program between 2020 and the time they complete the study protocol.

Study Design This will be a pre-test and post test quasi-experimental study for a duration of 12-weeks. When enrollment to participate is confirmed and informed consent is received , participants will complete the platform to evaluate athlete knowledge of sports nutrition questionnaire (PEAK-NQ), three factor eating questionnaire (TFEQ)-R18 (cognitive restraint eating subscale only), low energy availability male questionnaire (LEAM-Q) or low energy availability female questionnaire (LEAF-Q), a 5-day food intake journal food management questionnaire , athlete diet index questionnaire (ADI) , athlete food choice questionnaire (AFCQ) , surface anthropometry , resting metabolic rate assessment , dual-energy x-ray absorptiometry (DXA) scan for bone mineral content and body composition, and DXA bone mineral density (regional). All measurements will be repeated on week 12 (final) to complete the assessment.

The project will be staged at the Institut National du Sport du Québec. It is a national multisport training and sport science/medical service institute for more than 10 national elite sport programs.

MEASUREMENTS AND STUDY INSTRUMENTS

Surface Anthropometry Anthropometric profiles, including body mass, standing height, bone breadths at 6 sites, girths at 5 sites and skinfolds at eight sites will be measured by a level III accredited anthropometrist from the International Society for the Advancement of Kinanthropometry (ISAK) with a technical error of measurement of ≤ 2.0% for sum of eight skinfolds and ≤ 1.0% for all other measures. All measurements will be made on the right side of the body using ISAK techniques previously described (Stewart et al., 2011). Standing height will be measured using a stadiometer (Rosscraft, Surrey, BC, Canada), body mass on a calibrated digital scale with a precision of ± 0.1 kg (BWB-800S Tanita, Illinois, USA), girths with a flexible steel measuring tape (Rosscraft, Surey, BC, Canada), bone breadth with small bone caliper (Rosscraft, Surrey, BC, Canada) and skinfolds with a Harpenden calipers (Baty International, Burgess Hill, England).

The calculations of phantom z score of bone breadths and girths, body mass index, lean mass index and anthropometric somatotype will be performed as previously described (Norton and Olds, 1996 & Slater et al., 2006).

Dual-Energy x-Ray Absorptiometry Scanner To minimize biological variability, scans will be conducted in an overnight fasted (≥8 hours post-prandial), rested state following a low training volume day. Participants will be instructed to maintain their usual dietary habits the day prior to testing, with the addition of 500ml of water at each eating occasion. To confirm hydration status, specific gravity of the first void urine sample on the morning of testing will be assessed using an automated refractometer (Atago 4410 Digital Urine Refractometer, Tokyo, Japan).

The DXA (Lunar Prodigy, GE Healthcare, Madison, WI) will be calibrated with phantoms as per manufacturer guidelines each day before measurement. All scans will be conducted by the same bone densitometry technologist, certified through the International Society of Bone Densitometry. The USA (Combined NHANES (ages 20-30) / Lunar (ages 20-40)) Total Body Reference Population (v113) will be used as the reference database with analysis performed using GE Encore version 13.60 software (GE, Madison, WI). The thickness mode will be determined by the auto scan feature in the software and we will adhere to all safety protocols as per the institution's radiation safety protection plan.

DXA Scanning Protocol for Body Composition Participants will be asked to wear minimal clothing without metal zippers, tags, or studs and with all metal jewelry removed. Participants will be positioned according to protocols previously described (Nana et al., 2015). Participants too tall to fit within the defined scanning area will undertake two scans. The first scan captured the body from the inferior mandibular edge while the head was in the Frankfurt plane. After body repositioning and realigning the head in the Frankfurt plane, the second scan will capture the inferior mandibular edge to the vertex of the head. The results will be combined post analysis to estimate whole body fat mass, lean body mass, fat free mass and visceral adipose tissue. All scans will be analyzed automatically by the DXA software, but all regions of interest will be reconfirmed by the technician before being included in the subsequent statistical analysis. Fat-free and fat mass indexes will be calculated as previously described (Vanltallie et al., 1990).

DXA Scanning Protocol for Bone Mineral Content (BMD) Regional BMD will be determined according to standard positioning protocol from the International Society for Clinical Densitometry (ISCD Official Positions-Adults 2019). Measures will include BMD of the left and right hip, left and right radius and anterior-posterior lumbar spine. BMD age and ethnicity matched z-score estimated by the software will be used to identify low BMD values (z-score < -1) (Mountjoy et al., 2018).

Blood Samples All participants will provide blood samples after an overnight fast (≥8 hours post-prandial), which will be analyzed for complete blood cell count, calcidiol, RBC magnesium, vitamin B12, ferritin, c-reactive protein, glucose, insulin, lipids, ferritin, free-triiodothyronine (T3), leptin, cortisol, follicle-stimulating hormone (FSH) and luteinizing hormone (LH). All female participants will be analyzed for prolactin and 17-beta-estradiol (estradiol). All male participants will be analyzed for total-testosterone (total-TES), free-testosterone (free-TES) and sex hormone-binding globulin (SHBG). For consistency, all blood samples will be collected by a registered nurse at Institut National du Sport du Québec and analyzed externally by an accredited laboratory as per Institut National du Sport du Québec operational procedures.

Platform to Evaluate Athlete Knowledge of Sports Nutrition Questionnaire (PEAK-NQ) Athlete knowledge on sport nutrition will be assessed through a validated 50-item electronic questionnaire (Tam et al., 2021). It will be based on a total score of 75 across two sections: General Nutrition and Sports Nutrition. Correct answers are given one mark. Incorrect and "not sure" responses are given a zero mark. The items with multiple correct answers will score one mark per correct answer and be deducted one mark per incorrect option. Negative scores resulting from multiple incorrect answers will be adjusted to zero.

Athlete Food Choice Questionnaire (AFCQ) To account for factors that reportedly influence food choices in elite athletes will be assessed by the AFCQ. It is a validated 32-items questionnaire to assess 9-factors influencing food choices in elite athletes (Thurecht et al., 2021). Items will be presented as neutral statements and participants rank each on a frequency scale from 1 (never) to 5 (always). Food choice will be referred to foods and beverages.

Athlete Diet Index (ADI) The participants eating habits will be assess with the ADI questionnaire. It is a food frequency questionnaire based on reported habits over the last 7 days and was validated in elite athletes across multiple sport disciplines (Capling et al, 2021). A total score (out of a possible 125) will be calculated from the sum of the individual sub-scores; with a higher score indicating greater compliance with dietary recommendations for healthy and sport performance/recovery. The total ADI score, sub-scores, and non-scored information (ie: 7 day training log, dietary supplement use) will be used in combination to provide an indication of overall diet quality and dietary patterns of the athletes. Although the sub-score for healthy eating are based on the Australian guidelines to healthy eating, the principals are similar to the Canadian Food Guide and will therefore be included in the group analysis (Government of Canada, n.d. & and Australian Government, n.d.)

Dietary Intake Journal Each athlete will complete a 5-consecutive day dietary intake report within the week while using the Keenoa (Montréal, Québec, Canada) phone application (Ji et al, 2020). The intake assessment will include a day of rest, and 4 days of coach directed training. Athletes will receive detailed online instructions on how to record all food, fluid and dietary supplement intake. During this investigation, the researcher will use the participant's email to send an invitation to download the app on their smartphone, which will connect the user to the PhD candidate. Participants will be asked to weigh and take pictures of each food item with their smartphone prior to consumption. A food scale will be provided to facilitate data capture. If the app recognizes the food item(s), it will display selected options for the users to confirm the right identity of the food. Items could range from a single item (ie: apple) to composite items (ie: lasagna). Alternatively, participants could search and record food items manually from a database linked to the Canadian Nutrient File (2015). If the athlete ate out or is unable to find a suitable food match among the available choices on the app, they will be instructed to provide the name of the restaurant food, and fluid orders with size; or name of the food with brand and portion size, respectively, to enable cross-checking. The PhD candidate will review all dietary records and analysis reports for consistency.

Food Management Questionnaire This non-validated questionnaire will be used to describe some basic factors associated with the athlete's capability based on the COM-B model to manage food and fluid availability and preparation for oral consumption during the training week. It is divided into 3 main subcategories such as culinary environment at his/her place of residence, food availability and food preparation.

Low energy availability male questionnaire (LEAM-Q) Participants will complete a 42-item questionnaire to screen for self-reported physiological symptoms related to low energy availability (Lundy et al., 2022). Higher total scores indicate a higher relative risk of low energy availability, but with a lower sex-drive being a more sensitive indicator. Low sex drive is identified when 2 or more score on A1 or 2 or more is scored on B1 and 1 or more on B2.

Low Energy Availability in Females Questionnaire (LEAF-Q) Female participants will complete a 25-item questionnaire to screen for self-reported physiological symptoms related to low energy availability (Melin et al., 2014). Participants will be subsequently categorized as being at risk for the RED-S if their total score is ≥8.

Eating Disorder Examination Questionnaire (EDE-Q 6.0) All participants will complete a 28-item questionnaire derived from the semi-structured interview Eating Disorder Examination to assess the range and severity of features associated with a diagnosis of eating disorder using 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and a global score (Fairburn et al, 2008). It focuses on the past 28 days and uses a seven-point rating scale (0-6). Total score > 2.5 to ensure vulnerable subgroups are not subjected to mental health triggers that may encourage problems with eating (Kuikman et al., 2021). The 2 subscales related to shape and weight concerns will be used at pre and post testing to assess change in self-reported concerns with physique.

Three Factor Eating Questionnaire R18 (TFEQ-R18) The TFEQ-R18 refers to current dietary practice and measures 3 different aspects of eating behavior: restrained eating (conscious restriction of food intake to control body weight or to promote weight loss), uncontrolled eating (tendency to eat more than usual due to a loss of control over intake accompanied by subjective feelings of hunger), and emotional eating (inability to resist emotional cues) (de Lauzon et al., 2004). The questionnaire consists of 18 items on a 4-point response scale and items are scored, summated and transformed into a 0-100 scale for each behaviour as previously described. Higher scores in the respective scales indicate greater cognitive restraint, uncontrolled, or emotional eating. For the purpose of this investigation, the questions for calculating the cognitive restraint eating behaviours score will only be used at each testing time point to characterize restraint eating. The TFEQ-R18 restraint eating score (questions 2, 11, 12, 15, 16 and 18) was selected over EDE-Q 6.0 restraint eating score because it has been associated with athletes at risk of LEA/RED-S as well as surrogate markers of LEA in the athletic population (Jurov et al., 2021, Viner et al., 2015 and Sesbreno et al., 2023).

Measured Resting Metabolic Rate Measured resting metabolic rate (RMR) will be measured, in a fasting state, to operate the Goldberg cut-off to assess cases of over- or under-reporting as previously described as well as to calculate the measured:predicted RMR ratio for LEA screening (Black, 2000 and Mountjoy et al., 2018). Whole body mRMR and substrate utilisation were determined from the rates of oxygen consumption (VO2) and carbon dioxide production (VCO2), measured using a flow-through open circuit respirometry system with a ventilated hood (Field Metabolic System, Sable Systems International, Las Vegas, NV). The rates of VO2 and VCO2 production were calculated using equations previously described and adapted for its application with a ventilated hood (Brown et al., 1984). This approach allowed for a constant measurement and subsequent correction for the dilution effect of water vapor pressure on VO2 and VCO2. A background baselining technique was then applied to correct for analyzer drift and changes in environmental conditions. Substrate utilisation and their caloric equivalents were calculated as described previously (Péronnet et al., 1991). This could be scheduled within 2 weeks after fasted bloodwork if flexibility is required for your schedule.

Low Energy Availability in Females Questionnaire (LEAF-Q) Female participants will complete a 25-item questionnaire to screen for self-reported physiological symptoms related to low energy availability (Melin et al., 2014). Participants will be subsequently categorized as being at risk for the RED-S if their total score is ≥8.

Low energy availability male questionnaire (LEAM-Q) Participants will complete a 42-item questionnaire to screen for self-reported physiological symptoms related to low energy availability (Lundy et al., 2022). Higher total scores indicate a higher relative risk of low energy availability, but with a lower sex-drive being a more sensitive indicator. Low sex drive is identified when 2 or more score on A1 or 2 or more is scored on B1 and 1 or more on B2.

Indicators of Low Energy Availability (LEA) The primary indicators of LEA in all participants will be defined as low BMD z-score <-1.0 (Mountjoy et al., 2018). For female participants, a primary indicator will also consist of amenorrhea, defined as the absence of menstrual period for at least three consecutive months; a LEAF-Q score≥8; and in the absence of oral contraceptive agents, low estradiol, FSH, and LH, according to phase of the menstrual cycle as previously reported (Melin et al. 2015). For male participants, a primary indicator will also consist of low free- and total testosterone (lower quartile of normal range) as previously reported (Stenqvist et al., 2021 & Tenforde et al., 2016). Secondary indicators of LEA will be selected based on previous studies reporting signs of surrogate markers of LEA in male and female athletes that include glucose, free-triiodothyronine, low-density lipoprotein cholesterol, insulin, and leptin (Sesbreno et al., 2022a, in preparation; Stenqvist et al., 2021, Sygo et al., 2018).

Treatment Schedule and Documentation During week 1 of the observational period, all participants will be scheduled to receive individualized counselling in nutrition by a registered dietitian employed at l'Institut National du Sport du Québec (INS Québec) with field expertise in sport nutrition in high performance sports. The initial meeting will involve a comprehensive nutrition assessment with information gathered during the pre-assessment period (week 0) of the study protocol. The assessment will inform key dietary prioritize based on sport/training and medical objectives/requirements and recommendations and dietary plans will be developed and shared with the athlete to inform eating habits. Follow up appointments over the 11 week observation will be mutually developed and agreed upon between athlete and dietitian, unless a referral is issued by a member of the medical and integrative support staff (coaches, strength & conditioning, physiotherapist, mental health professional, physiologist, etc..) team in agreement with the athlete.

During the initial and subsequent follow-up meetings, the athlete will complete the AFCQ on the day of the meeting before seeing the dietitian. The dietitian will be blinded to the responses in order to not influence the outcome of the appointment. The AFCQ is a novel tool is not yet used regularly in the Canadian high performance sport environment. The responses will be examined during the study analysis phase. At the end of each appointment, the dietitian will complete a SOAP (subjective/objective data, assessment and plan) note and the interventions listed under plans will include a code based on electronic nutrition care process (NCP) terminology (https://www.ncpro.org/modules/portal/publications.cfm) for greater clarity. Subsequently, the participant's alpha numeric ID, date of intervention and plan section of the SOAP note, which includes the written intervention and NCP intervention code will be shared with two members of the research team (who are registered sport/research dietitians) who will never be directly implicated in the data collection, assessment and development of plans to manage athletes participating in the study. Their specific role will be to independently code the registered dietitians SOAP note intervention based on the Behaviour Change Term Taxonomy (http://www.behaviourchangewheel.com/about-wheel) for analysis accordingly to the Capacity Opportunity Motivation-Behaviour Change (COM-B) model. The code will not be accepted into the database until independent agreement is reached. After 3 failed attempts, a third researcher (who is a registered sport/research dietitian) will independently code the intervention. In this case, the popular vote will determine the coding of the intervention for inclusion in the database for analysis. All registered dietitians involved in the project for delivering care to the athlete will complete all online tutorials for the NCP intervention coding whereas and those not involved in care, but only in coding the professional's interventions for project analysis will complete tutorials for both the NCP intervention and Behaviour Change Term Taxonomy (BCT) coding for quality assurance (https://www.ncpro.org/encpt-tutorials).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Active to participate in training and competition
* Able-bodied sport program
* Having given informed consent

Exclusion Criteria:

* Eating Disorder Examination Questionnaire 6.0 total score > 2.50 (women) and > 1.68 (male)
* Unable to understand spoken and written English

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Nutrition knowledge | 12 weeks
  PEAK-NQ
Change in carbohydrate intake | 12 weeks
  Food Record

SECONDARY OUTCOMES:
Change in food frequency intake of carbohydrate rich foods | 12 weeks
  Athlete Diet Index

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided